CLINICAL TRIAL: NCT04399512
Title: Evaluation of Oral Health Status in Patients With Cirrhosis and Effect of Dental Treatment on MELD Score of Cirrhosis Patients
Brief Title: Oral Health Status in Patients With Cirrhosis and Effect of Dental Treatment on MELD Score of Cirrhosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: swatiendo18787
Record Dates: First submitted 2020-04-24; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2019-12

CONDITIONS: Liver Cirrhosis; Periapical Lesions
Keywords: Apical periodontitis; liver disease; root canal treatment
MeSH Terms: conditions — Liver Cirrhosis; Periapical Periodontitis; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Cross-sectional and Interventional study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with liver cirrhosis (Active Comparator): prevalence of apical periodontitis will be checked and non-surgical root canal treatment will be given to the patients with apical periodontitis and change in MELD(model for end stage liver disease) will be checked after treatment.
  Interventions: Procedure: Nonsurgical root canal treatment
- Normal healthy patients (Active Comparator): prevalence of apical periodontitis will be checked and non-surgical root canal treatment will be given to the patients with apical periodontitis
  Interventions: Procedure: Nonsurgical root canal treatment

INTERVENTIONS:
Procedure: Nonsurgical root canal treatment — Nonsurgical root canal treatment will be given

SUMMARY:
It has been found that there is an association between prevalence of odontogenic infection and systemic diseases.Cirrhosis has also been associated with poor oral health status.Treating those patients accordingly can help in reducing the source of infection to some extent and may be associated with reduction in mortality.

DETAILED DESCRIPTION:
Patients will be selected according to inclusion and exclusion criteria.Written informed consent will be taken from each participant after being informed about study .There will be two groups1) cirrhosis patients 2)normal healthy patients.Prevalence of apical periodontitis will be measured in both groups by intraoral examination,digital panoramic radiography.. MELD score will be recorded in cirrhosis patients at this stage.Non surgical root canal treatment will be performed in teeth with apical periodontitis. Periapical healing will be checked with the help of PAI Score given by Orstavik. In Cirrhosis patients MELD Score will be measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria:(cirrhosis patients)

1. Known patient of cirrhosis(Diagnosis of cirrhosis is based on blood testing, medical imaging, and liver biopsy.) with mature permanent teeth .
2. Age35-55 years
3. > or equal to 8 natural teeth(excluding 3rd molars);
4. I.N.R < 3.5

   -

Exclusion Criteria:(Cirrhosis patients)

1. Patient having systemic disorders other than hepatic disease(e.g. HIV, osteoporosis,diabetes,cardiovascular disease)
2. Pregnancy
3. Use of systemic and topical antibiotic treatment within 3 months prior to the start of the study.

The eligibility criteria of the control group were the same for the cirrhosis group, except for the presence of liver disease. Cirrhosis patients were matched with controls according to sex, age (± 3 years old) and current smoking status and alcohol satus (yes/no).

-

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
prevalence of apical periodontitis in patients with cirrhosis and healthy patients. | Baseline to 12 months
  periapical index score will be assigned to intraoral periapical radiograph of teeth showing periapical radiolucency in orthopantomogram of each patient .PAI score 3,4,5 will be diagnosed with apical periodontitis .
  Score Description
  1. Normal periapical structure
  2. Small changes in bone structure
  3. Changes in bone structure with some mineral loss
  4. Periodontitis with well-defined radiolucent area
  5. Severe periodontitis with exacerbating features

SECONDARY OUTCOMES:
association of prevalence of marginal and apical periodontitis with mortality measured by MELD score in cirrhosis patients | Baseline to 12 months
  Model for end stage liver disease score of all cirrhotic patients will be calculated using serum bilirubin, serum creatinine, and International Normalized Ratio (INR) by the formula 9.57 × loge (creatinine) + 3.78 × loge (total bilirubin) + 11.2 × loge (INR) + 6.43.
Clinical and radiographic success | Baseline to 12 months
  Clinical success will be assessed by absence of clinical signs and symptoms and radiographically PAI score 1 ,2 will be considered as healed.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India